CLINICAL TRIAL: NCT04082572
Title: Neoadjuvant Pembrolizumab for Patients With Mismatch Repair Deficient Locally Advanced Solid Cancers
Brief Title: Pembrolizumab Before Surgery for the Treatment of Mismatch Repair Deficient Locally Advanced Solid Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1182; NCI-2019-05822 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1182 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Malignant Solid Neoplasm
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for 1 year in the absence of disease progression or unacceptable toxicity. Patients who do not respond to pembrolizumab and stop the treatment after 2 doses may undergo surgery within 6 months.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works before surgery in treating patients with mismatch repair deficient solid cancers that have spread to nearby tissue or lymph nodes (locally advanced). Cancer is caused by changes (mutations) to genes (DNA) that control the way cells function, and some of these mutations can cause tumor cells to grow quickly and out of control. Microsatellite instability-high (MSI-H) tumors are made up of cancer cells that have a greater than normal number of genetic markers called microsatellites. These cancers may have defects in the ability to correct mutations that occur when DNA is copied in the cell. Similarly, mismatch repair deficient tumors (dMMR) may have difficulty repairing some type of genetic mutation during cellular replication that may affect tumor's response to cancer therapy. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of neo-adjuvant pembrolizumab in patients with locally advanced (unresectable primary cancer or resectable primary cancer with a high chance of recurrence) mismatch repair protein deficiency (dMMR) solid organ tumors by Common Terminology Criteria for Adverse Events (CTCAE) assessed toxicity and post-surgical complication assessment by the Clavien-Dindo classification.

II. To assess the rate of complete pathological response for patients who undergo surgical resection following at least 3 doses of neoadjuvant pembrolizumab.

SECONDARY OBJECTIVES:

I. To quantify the rate of organ sparing at 1 year for all patients treated with one dose of pembrolizumab (intent to treat) and those patients who receive at least 3 doses of neoadjuvant pembrolizumab and decline to undergo surgical resection and opt to continue receiving pembrolizumab for a total of 1 year.

II. To assess radiographic tumor response to neoadjuvant pembrolizumab. III. To estimate the relapse-free survival and overall survival in all enrolled participants.

IV. To determine the overall rates of pathological response to neoadjuvant pembrolizumab.

V. To assess the rate of complete pathological response (intent to treat) for patients who undergo surgical resection following at least 1 dose of neoadjuvant pembrolizumab.

EXPLORATORY OBJECTIVE:

I. To explore the predictive ability of changes in circulating tumor-derived deoxyriboucleic acid (ctDNA) for efficacy endpoints.

II. To determine if total mutational burden correlate with response and extent of benefit from pembrolizumab.

III. To correlate pre-treatment tumor samples tumor-immune microenvironment (for example Teffector cell populations; CD4 subsets; T-regulatory populations; B cell populations; dendritic and macrophage populations) with efficacy endpoints.

IV. To compare targeted gene expression profiles of immune related genes and genes pertaining to common cancer signaling pathways in pre-treatment samples and also the change in these factors for cases with both pre and on-treatment (i.e. at time of resection) tumor samples of responders (stable disease or radiographic response prior to resection) versus non-responders (progression prior to resection).

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days for 1 year in the absence of disease progression or unacceptable toxicity. Patients who do not respond to pembrolizumab and stop the treatment after 2 doses may undergo surgery within 6 months.

After completion of study treatment, patients are followed up at 30 days, every 6 weeks for 1 year, every 9-12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of solid cancer
* Solid cancer that is deficient in mismatch repair (dMMR) or microsatellite instability high (MSI-H) as determined by one of three methods:

  * Immunohistochemistry determined dMMR by complete loss of MLH1, PMS2, MSH2 or MSH6
  * Polymerase chain reaction (PCR) determined microsatellite instability at > 30% of tested microsatellites
  * Next-generation sequencing determined MSI-H based upon instability at multiple microsatellites as determined by the specific next generation sequencing panel
* Locally advanced cancer defined as either an unresectable primary cancer or a resectable primary cancer with a high chance of recurrence (defined as an estimated greater or equal to 20% chance of recurrence by the treating physician). A resectable primary may include locoregional disease, as long as all disease is felt by the treating physician to be in a resectable distribution
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 (unless discussed and approved by study principal investigator [PI])
* Have available archival tumor tissue. Availability will be met as long as a request to obtain formalin-fixed, paraffin embedded (FFPE) tissue blocks (preferred) or slides has been made (unless discussed and approved by study PI)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of signing study consent
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least (120 days [corresponding to time needed to eliminate any study treatment(s) plus 30 days (a menstruation cycle) for risk of genotoxicity]) after the last dose of study treatment
* Absolute neutrophil count (ANC) >= 1500/uL (within 14 days prior to the start of study treatment)
* Platelets >= 100 000/uL (within 14 days prior to the start of study treatment)
* Hemoglobin >= 8.0 g/dL or >= 5.6 mmol/L (within 14 days prior to the start of study treatment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (within 14 days prior to the start of study treatment)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (within 14 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases) (within 14 days prior to the start of study treatment)
* International normalized ratio (INR) OR prothrombin time (PT) activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (within 14 days prior to the start of study treatment)

Exclusion Criteria:

* A woman of childbearing potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137)
* Has received prior systemic anti-cancer therapy including investigational agents within 2 weeks of study treatment. Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible
* If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has a known additional malignancy that is progressing or has required active treatment within the past 1 year. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) or other similar good prognosis cancer with recurrence rates expected to be < 10% that have undergone potentially curative therapy are not excluded
* Known metastatic sites of disease. Note: locoregional lymph nodes or tumor deposits are not considered metastatic disease
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV)
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection. Note: no testing for hepatitis B and hepatitis C is required unless mandated by local health authority
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Overman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ludford K, Ho WJ, Thomas JV, Raghav KPS, Murphy MB, Fleming ND, Lee MS, Smaglo BG, You YN, Tillman MM, Kamiya-Matsuoka C, Thirumurthi S, Messick C, Johnson B, Vilar E, Dasari A, Shin S, Hernandez A, Yuan X, Yang H, Foo WC, Qiao W, Maru D, Kopetz S, Overman MJ. Neoadjuvant Pembrolizumab in Localized Microsatellite Instability High/Deficient Mismatch Repair Solid Tumors. J Clin Oncol. 2023 Apr 20;41(12):2181-2190. doi: 10.1200/JCO.22.01351. Epub 2023 Jan 9. PMID 36623241
- [Derived] Mendonca Gorgulho C, Krishnamurthy A, Lanzi A, Galon J, Housseau F, Kaneno R, Lotze MT. Gutting it Out: Developing Effective Immunotherapies for Patients With Colorectal Cancer. J Immunother. 2021 Feb-Mar 01;44(2):49-62. doi: 10.1097/CJI.0000000000000357. PMID 33416261
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October 31, 2019, and March 25, 2021
Groups:
- Neoadjuvant Pembrolizumab in Localized MSI Instability High/Deficient Mismatch Repair Solid Tumors: Pembrolizumab given pre-operatively for 6 months in patients with locally advanced (unresectable primary cancer or a resectable primary cancer with a high chance of recurrence) dMMR solid organ tumors
Period: Overall Study
Arm/Group | Neoadjuvant Pembrolizumab in Localized MSI Instability High/Deficient Mismatch Repair Solid Tumors
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Pembrolizumab in Localized MSI Instability High/Deficient Mismatch Repair Solid Tumors
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 62 [25 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR).
Description: Number of patients with Pathologic complete response (pCR) as defined by absence of any residual viable tumor of the macroscopically identifiable tumor bed or lymph node after 3 doses.
Time Frame: 1 year
Population: 35 patients were enrolled in the study. The primary efficacy end point was evaluable in only 15 patients. 17 patients (49%) had surgical resection. However, 2 patients had a resection after 1 and 2 cycles of treatment. Thus only 15 patients were found to be eligible (resection after 3 cycles of treatment with pembrolizumab).
Measure: Number; unit: Percentage
Arm/Group | Neoadjuvant Pembrolizumab in Localized MSI Instability High/Deficient Mismatch Repair Solid Tumors
Number analyzed (Participants) | 15
Percentage | 67

2. Primary Outcome: Safety of Neo-adjuvant Pembrolizumab in Patients With Locally Advanced (Unresectable Primary Cancer or Resectable Primary Cancer With a High Chance of Recurrence) Mismatch Repair Protein Deficiency (dMMR) Solid Organ Tumors.
Description: Number of patients that developed toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.
Time Frame: At 1 year
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Pembrolizumab in Localized MSI Instability High/Deficient Mismatch Repair Solid Tumors
Number analyzed (Participants) | 35
participants | 35

3. Primary Outcome: Post-surgical Complication Assessment by the Clavien- Dindo Classification.
Description: Number of patients with post surgical complication based on the Clavien-Dindo Classification
Time Frame: Up to 2 years
Population: 35 patients were enrolled in the study. Only 17 patients underwent resection. out of the 17 patients that underwent resection, 3 patients developed post surgical complications.
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Pembrolizumab in Localized MSI Instability High/Deficient Mismatch Repair Solid Tumors
Number analyzed (Participants) | 17
participants | 3

4. Secondary Outcome: Overall Response Rate
Description: The ORR was estimated using Recist 1.1. ORR (Complete response + Partial response)
Time Frame: From treatment start till death or last follow-up, assessed up to 2 years
Population: 35 patients were enrolled but only 33 patients were evaluable for radiographic response. 2 patients were not evaluable due to clinical progression and death due to an unrelated hip fracture in a 90 year old patient before restaging.
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Pembrolizumab in Localized MSI Instability High/Deficient Mismatch Repair Solid Tumors
Number analyzed (Participants) | 33
participants | 27

5. Secondary Outcome: Radiographic Tumor Response to Neoadjuvant Pembrolizumab.
Description: Best overall RECIST response as determined by the number of patients with Partial Response and or Complete Response measured using Recist v1.1
Time Frame: 1 year
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Pembrolizumab in Localized MSI Instability High/Deficient Mismatch Repair Solid Tumors
Number analyzed (Participants) | 33
participants | 27

ADVERSE EVENTS:
Time Frame: 2 Year
Groups:
- Neoadjuvant Pembrolizumab in Localized MSI Instability High/Deficient Mismatch Repair Solid Tumors: Pembrolizumab
Arm/Group | Neoadjuvant Pembrolizumab in Localized MSI Instability High/Deficient Mismatch Repair Solid Tumors
All-Cause Mortality (participants affected / at risk) | 2/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 35/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Pembrolizumab in Localized MSI Instability High/Deficient Mismatch Repair Solid Tumors (N=35)
Anemia (Blood and lymphatic system disorders) | 31
Sinus Tachycardia (Cardiac disorders) | 4
Sinus bradycardia (Cardiac disorders) | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Hearing impaired (Nervous system disorders) | 1
Hypothyroidism (Endocrine disorders) | 4
Hypoparathyroidism (Endocrine disorders) | 1
Hyperthryroidism (Endocrine disorders) | 2
Blurred Vision (Eye disorders) | 3
Watering Eyes (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 9
Anal hemorrhage (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Rectal hemorrhage (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 7
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Pain (General disorders) | 1
Sepsis (Infections and infestations) | 2
Urinary Tract Infection (Renal and urinary disorders) | 2
Vulval Infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 14
Alkaline phosphatase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 5
Investigations - Other, specify (Investigations) | 27
Neutrophil count decreased (Investigations) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 1
Hypercalcemia (Investigations) | 3
Hyperglycemia (Investigations) | 20
Hyperkalemia (Investigations) | 3
Hypermagnesemia (Investigations) | 1
Hyperuricemia (Investigations) | 11
Hypoalbuminemia (Investigations) | 1
Hypokalemia (Investigations) | 7
Hypomagnesemia (Investigations) | 1
Hyponatremia (Investigations) | 8
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Memory impairment (Nervous system disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Insomnia (Nervous system disorders) | 1
Urinary Urgency (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Vaginal Pain (Reproductive system and breast disorders) | 1
Uterine Hemorrahage (Reproductive system and breast disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1
Vascular disorders - Other, specif (Vascular disorders) | 1
Hot flashes (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT04082572/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT04082572/ICF_000.pdf